**Title:** Study 3 Learning Verbs and Pronouns

NCT Number: NCT05193500

**Document date**: 10/20/2020

#### Parental Permission Form for Minors, IRB-FY2018-2041

Your child has been invited to take part in a research study to learn more about how children learn to understand language. This study will be conducted by Dr. Sudha Arunachalam of the Communicative Sciences and Disorders department at the Steinhardt School of Culture, Education, and Human Development, New York University, and Dr. Rhiannon Luyster of the Communicative Sciences and Disorders department at Emerson College.

If you give permission for your child's participation in this study, your child will be asked to play some games with an experimenter on your computer or tablet via Zoom videoconferencing software. You will be with your child the entire time.

Your child will be audio and video recorded. You and your child may review these recordings and request that all or any portion of the recordings be destroyed.

Participation in this study will involve approximately 1 hour of your child's time. We intend to enroll 400 children in the study,

Participation in this study is voluntary. Your child may refuse to participate or withdraw at any time without penalty. Please read the rest of this parental permission form for more information about the study.

#### **Risks and Discomfort**

Your child may get tired or restless during the tasks. You can take a break at any time, and can stop early at your discretion.

The main risk of allowing us to use and store your information for research is a potential loss of privacy. We will protect your privacy by labeling your information with a code rather than your or your child's name, and keeping the key to the code in a password-protected computer. For videoconferencing parts of the study, the experimenter will provide private access to your Zoom meeting and store the meeting recording on a secure database in a password-protected file.

There may be unforeseen risks to the study. If new risks are identified the study staff will update you in a timely way about any new information that might affect you or your child's health, welfare, or decision to participate.

### **Benefits**

Although your child will receive no direct benefits, this research may help the investigator understand how children learn language. This information may be used to inform future research about how to help children learn language.

# Compensation

There is no compensation for your participation. Your participation along with your child will be compensated as described in the other consent form.



## Confidentiality

Confidentiality of your child's research records will be strictly maintained. Any identifiable data that is collected from you or your child will be identified by a study ID. Only the researchers will have access to the master-code that links you and your child's personal information to the study ID number. The researchers will store the research data in locked files and a password-protected computer, and it will be backed up on a password-protected internet archive database. The data will only be accessible to the researchers. The signed consent forms will be kept separate from the research data.

Information derived from this study will be used for research purposes, which may involve publication and teaching. Your and your child's information may be used in publications or presentations. However, the information will not include any personal information that will allow either of you to be identified. Any reports of the data will emphasize group patterns rather than individual performance. If your child's individual results are discussed, your child's identity will be protected by using a study ID number rather than names or other identifying information. In every case, anonymity is strictly preserved.

Information not containing identifiers may be used in future research or shared with other researchers without your additional permission or your child's additional consent.

A description of this clinical trial will be available on http://www.ClinicalTrials.gov as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

Clinically Relevant Data The following results from this study may be clinically relevant to your child: scores on standardized assessments of language and cognition. You will receive these results if you choose. However, although the assessments are standard, your child did not undertake them for clinical purposes in a clinical setting, and the scores therefore may not have any relevance in providing clinical or medical treatment for your child. Our study staff will not be able to provide an interpretation of the results. We suggest that you bring these scores to your child's pediatrician or other professional, who may be able to decide if the assessments are helpful in providing care for your child.

### **Voluntary Nature of Participation**

Participation in this study is voluntary. Your child may refuse to participate or withdraw at any time without penalty. Your child has the right to skip or not answer any questions he/she/they prefer not to answer.

Nonparticipation or withdrawal will not affect any services you or your child receives at the NYU Speech-Language-Hearing Clinic or Emerson College.

# **Contact Information**

If there is anything about the study or your child's participation that is unclear or that you do not understand, or if you have questions or wish to report a research-related problem, you may contact Dr. Sudha Arunachalam at (212) 998-5230 or <a href="sudha@nyu.edu">sudha@nyu.edu</a>, or Dr. Rhiannon Luyster at rhiannon luyster@emerson.edu or (617) 824-3503.



If you have any questions about your child's rights as a research subject or complaints regarding this research study, or you are unable to reach the research staff, you may contact a person independent of the research team at the Biomedical Research Alliance of New York Institutional Review Board at 516-318-6877. Questions, concerns or complaints about research can also be registered with the Biomedical Research Alliance of New York Institutional Review Board at <a href="https://www.branyirb.com/concerns-about-research">www.branyirb.com/concerns-about-research</a>

| Permission for Child to Participate | |
|---|---|
| Name of Child | |
| | <del></del> |
| Parent's Signature | Date |
| Participating in future research | |
| Are you interested in participating in future research wit you to participation. We will simply contact you when we enjoy, and ask if you are interested in participating at the | e have another study that we think your child may |
| ☐ Yes, you may contact me about additional research | opportunities <b>online only</b> . |